CLINICAL TRIAL: NCT05269069
Title: Impact of Rheumatoid Arthritis on Body Composition, Bone Marrow Adiposity and Bone Mineral Density: a Case-control Study
Acronym: RAFAT
Status: Terminated | Type: Observational
Why Stopped: The sponsor decided to stop financing the study.
Sponsor: University Hospital, Lille (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021_0845; 2021-A03187-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-02-07; First posted 2022-03-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Body composition; rheumatoid arthritis; visceral adiposity; marrow adiposity; bone mineral density
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with rheumatoid arthritis: patients with rheumatoid arthritis
  Interventions: Other: Assessment of body composition, bone mineral density and bone marrow adiposity.
- Control group: healthy volunteers without rheumatoid arthritis matched for age, sex, BMI and menopausal status
  Interventions: Other: Assessment of body composition, bone mineral density and bone marrow adiposity.

INTERVENTIONS:
Other: Assessment of body composition, bone mineral density and bone marrow adiposity. — DXA for body composition and bone mineral density, MRI for bone marrow adiposity and blood tests (leptine, CTX, P1NP)

SUMMARY:
During rheumatoid arthritis (RA) (in comparison with control subjects), body composition is altered with a loss of lean body mass, bone mass and an accumulation of fat mass.

Determination of total body fat and particularly its abdominal distribution (visceral adiposity) is important because of the cardiovascular (excess cardiovascular risk), metabolic (insulin resistance, diabetes and dyslipidemia) and bone (increased fracture risk) risks associated with this endocrine organ. Moreover, we do not have data concerning medullary adiposity in RA.

This pilot case-control study will be compare body composition, bone marrow adiposity and bone mineral density in patients with RA versus healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Subjects:

Males and females of age (age ≥ 18 years). Patients with RA according to American College of Rheumatology/EULAR 2010 criteria, Patients who have signed the informed consent

Controls:

Males and females of age (age ≥ 18 years). subjects who have signed the informed consent

Exclusion Criteria:

* Patients who have received more than three anti-TNFinhibitors
* Patients who have previously received a Janus kinase (JAK) inhibitor
* Patients with concomitant therapies as described below :

A combination with methotrexate is allowed if methotrexate is started ≥3 months before the start of the study and at a stable dosage (≤25 mg/week) for ≥4 weeks.

A combination to conventional synthetic DMARDs (csDMARDs) other than methotrexate is not allowed within 4 weeks before and/or during the clinical trial

* Corticosteroid therapy >10mg/d prednisolone equivalent is not allowed
* Intra-articular injections of corticosteroids are allowed if their number is less than or equal to 4
* Intravenous corticosteroid infusions are not allowed
* Immunosuppressants other than methotrexate are not allowed
* History or discovery of an osteoporotic fracture AND/OR T-score ≤-3 if ≥50 years old AND/OR Z-score ≤-3 if <50 years old during the screening phase,
* Corticosteroid therapy ≥ 10mg/d prednisolone equivalent,
* Pathologies or treatments affecting bone metabolism (breast cancer with antiaromatase, digestive malabsorption, stomach cancer, primary hyperparathyroidism, uncontrolled hyperthyroidism...),
* History of radiotherapy on the lumbar spine or the hip studied,
* Patients undergoing hormone replacement therapy (HRT) or patients already under anti-osteoporotic treatment (bisphosphonates, strontium ranelate, teriparatide or denosumab) apart from calcium and/or vitamin D supplementation, Chronic renal failure with creatinine clearance (CKD-EPI formula) ≤ 30 ml/min,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis and controls
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Measurement of visceral adiposity (VAT) in cm² at inclusion. | Baseline
  A whole body composition acquisition by dual energy x-ray absorptiometry (DXA) will calculate visceral adiposity

SECONDARY OUTCOMES:
Measures of lean body mass (LBM) in kg | Baseline
Measures of total body fat (TBF) in % | Baseline
Bone mineral density (BMD) measurements (in mg/cm²) at the lumbar spine (L1-L4) and total non-dominant hip | Baseline
Measurements of bone remodeling markers (CTX and P1NP) | Baseline
Level of Leptin | Baseline
Measurement of bone marrow adiposity (in %) at the lumbar spine | Baseline
Short Physical Performance Battery (SPPB) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Guillaume LETARTOUILLY, MD, MSc, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Salengro - Chu Lille, Lille, France